CLINICAL TRIAL: NCT01129544
Title: Multi-site Phase I/II Trial Evaluating the Treatment of SCID-X1 Patients With Retrovirus-mediated Gene Transfer
Brief Title: Gene Transfer for Severe Combined Immunodeficiency, X-linked (SCID-X1) Using a Self-inactivating (SIN) Gammaretroviral Vector
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Williams (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, David Williams, Chief of the Division of Hematology/Oncology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND14067
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Severe combined immunodeficiency; SCID; XSCID; SCID-X1
MeSH Terms: conditions — Severe Combined Immunodeficiency; X-Linked Combined Immunodeficiency Diseases | interventions — Genetic Engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene Transfer (Experimental): open label single arm study
  Interventions: Biological: Gene transfer

INTERVENTIONS:
Biological: Gene transfer — Three procedures: 1) Bone marrow harvest from the patient's posterior iliac crests. 2.) Chemotherapy conditioning with Busulfan 3)One time infusion of patient's transduced bone marrow cells.

SUMMARY:
Researchers are working on ways to treat SCID patients who don't have a matched brother or sister. One of the goals is to avoid the problems that happen with stem cell transplant from parents and unrelated people, such as repeat transplants, incomplete cure of the immune system, exposure to chemotherapy, and graft versus host disease.

The idea behind gene transfer is to replace the broken gene by putting a piece of genetic material (DNA) that has the normal gene into the child's cells. Gene transfer can only be done if we know which gene is missing or broken in the patient. For SCID-X1, gene transfer has been done in the laboratory and in two previous clinical trials by inserting the normal gene into stem cells from bone marrow. The bone marrow is the "factory" inside the bones that creates blood and immune cells. So fixing the gene in the bone marrow stem cells should fix the immune problem, without giving chemotherapy and without risk of graft versus host disease, because the child's own cells are used, rather than another person's. Out of the 20 subjects enrolled in the two previous trials, 18 are alive with better immune systems after gene transfer. Two of the surviving subjects received gene corrected cells over 10 years ago.

Gene transfer is still research for two reasons. One is that not enough children have been studied to tell if the procedure is consistently successful. Of the 20 children enrolled in the previous two trials, one child did not have correction of the immune system, and died of complications after undergoing stem cell transplant. The second important reason why gene transfer is research is that we are still learning about the side effects of gene transfer and how to do gene transfer safely. In the last two trials, 5 children have experienced a serious side effect. These children developed leukemia related to the gene transfer itself. Leukemia is a cancer of the white blood cells, a condition where a few white blood cells grow out of control. Of these children, 4 of the 5 have received chemotherapy (medication to treat cancer) and are currently in remission (no leukemia can be found by sensitive testing), whereas one died of gene transfer-related leukemia.

DETAILED DESCRIPTION:
Severe combined immunodeficiencies (SCID) are a heterogeneous group of inherited disorders characterized by a profound reduction or absence of T lymphocyte function. They arise from a variety of molecular defects which affect lymphocyte development and function. The most common form of SCID is an X-linked form (SCID-X1) which accounts for 40-50% of all cases. SCID-X1 is caused by defects in the common cytokine receptor chain, which was originally identified as a component of the high affinity interleukin-2 receptor (IL-2RG), but is now known to be an essential component of the IL-4, -7, -9 -15, and -21 cytokine receptor complexes. Classic SCID-X1 has an extremely poor prognosis without treatment. Death usually occurs in the first year of life from infectious complications unless definitive treatment can be administered. Until the recent advent of somatic gene therapy, hematopoietic stem cell transplantation (HSCT) offered the only curative option for patients with any form of SCID. If a genotypically matched sibling donor is available, HSCT is a highly successful procedure. However a genotypically matched family donor is only available for approximately 30% of patients. For the remaining individuals, alternative donor transplants, principally from matched unrelated or haploidentical parental donors have been performed. These approaches are still problematic with toxicity from ablative therapy, graft-versus-host disease and incomplete lymphoid reconstitution. Recent gene transfer trials have documented the efficacy of gene transfer in this disease, albeit with toxicity related to insertional mutagenesis. A new generation of self-inactivating (SIN) vectors has been developed which lack all enhancer-promoter elements of the LTR U3 region and are also devoid of all gammaretroviral coding regions. A SIN vector expressing the IL-2RG gene, pSRS11.EFS.IL2RG.pre* has been developed and has shown a reduction in mutagenic potential compared to LTR configuration in non-clinical studies. The current study is a phase I/II trial of somatic gene therapy for patients with SCID-X1.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SCID-X1 based on immunophenotype (<200 CD3+ autologous T cells, and confirmed by DNA sequencing)

   AND
2. Lack an HLA identical (A, B, C, DR, DQ) related donor

AND either one of the following:

1. Patients in good clinical condition who do not have a readily available HLA identical (A,B,C,DR,DQ) unrelated donor (readily available defined as: a donor confirmed within 6 weeks of searching, with ability to transplant within 3 months of diagnosis).

2. Patients with an active, therapy-resistant infection or other medical conditions that significantly increase the risk of allogeneic transplant. Examples of "therapy-resistant infections that significantly increase the risk of allogeneic transplant" include but are not limited to:

1. interstitial pneumonia due to adenovirus or parainfluenzae virus.
2. protracted diarrhea requiring total parenteral nutrition.
3. disseminated BCG infection.
4. virus-induced lymphoproliferative disease.
5. any active opportunistic infection (eg, due to Pneumocystis jiroveci, cytomegalovirus,cryptosporidium) that does not improve on medical management.
6. active and progressive pulmonary disease requiring mechanic ventilation. Inclusion of patients with disease-related organ dysfunction is justified by the known poor outcome with standard treatment and the potential life-saving nature of the treatment proposed. Patients who are on high-dose steroids or other immunosuppressive agents will also be considered eligible, because use of these drugs is common in patients with SCID and maternal T cell engraftment or who present with severe interstitial lung disease. Use of immunosuppressive drugs does not affect efficacy of hematopoietic cell transplantation, and therefore should not affect efficacy of gene transfer.

Exclusion Criteria:

1. No available molecular diagnosis confirming SCID-X1.
2. Patients who have an available HLA-identical related donor.
3. Diagnosis of active malignant disease other than EBV-associated lymphoproliferative disease
4. Patients with evidence of infection with HIV-1
5. Previous gene transfer
6. Major (life-threatening) congenital anomalies. Examples of "major (life-threatening) congenital anomalies" include, but are not limited to: unrepaired cyanotic heart disease, hypoplastic lungs, anencephaly or other major CNS malformations, other severe non-repairable malformations of the gastrointestinal or genitourinary tracts that significantly impair organ function.
7. Other conditions which in the opinion of the P.I. or co-investigators, contra-indicate collection and/or infusion of transduced cells or indicate patient's inability to follow the protocol. These may include for example clinical ineligibility to receive anesthesia, severe deterioration of clinical condition of the patient after collection of bone marrow but before infusion of transduced cells, or documented refusal or inability of the family to return for scheduled visits. There may be other unforeseen rare circumstances that would result in exclusion of the patient, such as sudden loss of legal guardianship.

Although the presentation of the disease may be variable in type, the severity of the immunodeficiency is uniform. The gene transfer protocol will be instituted in the place of haploidentical transplant for those patients who do not have a matched family donor or in whom an unrelated donor transplant is not indicated for the reasons specified above. Apart from the gene transfer protocol, the patients will not undergo additional procedures that would not form part of an equivalent haploidentical transplantation regimen, and will not receive conditioning chemotherapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
CD3 cell count post transfusion | 6 Months Post Gene Transfer
  Immunological reconstitution defined as absolute CD3 cells of >300/μl and PHA stimulation index >15 at 6 months post infusion
Incidence of life-threatening adverse reactions related to the gene therapy procedure. | Up to 15 years post gene transfer
  Incidence of life-threatening adverse reactions related to the gene therapy procedure.

SECONDARY OUTCOMES:
Molecular characterization of gene transfer. | Up to 15 years post gene transfer
Ability to mount antibody responses to vaccination. | Within 18 Months post standard vaccination to tentanus
Normalization of nutritional status, growth, and development | Up to 15 years post gene transfer

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whangbo, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Mattel Children's Hospital - UCLA, Los Angeles, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Clarke EL, Connell AJ, Six E, Kadry NA, Abbas AA, Hwang Y, Everett JK, Hofstaedter CE, Marsh R, Armant M, Kelsen J, Notarangelo LD, Collman RG, Hacein-Bey-Abina S, Kohn DB, Cavazzana M, Fischer A, Williams DA, Pai SY, Bushman FD. T cell dynamics and response of the microbiota after gene therapy to treat X-linked severe combined immunodeficiency. Genome Med. 2018 Sep 28;10(1):70. doi: 10.1186/s13073-018-0580-z. PMID 30261899
- [Derived] Hacein-Bey-Abina S, Pai SY, Gaspar HB, Armant M, Berry CC, Blanche S, Bleesing J, Blondeau J, de Boer H, Buckland KF, Caccavelli L, Cros G, De Oliveira S, Fernandez KS, Guo D, Harris CE, Hopkins G, Lehmann LE, Lim A, London WB, van der Loo JC, Malani N, Male F, Malik P, Marinovic MA, McNicol AM, Moshous D, Neven B, Oleastro M, Picard C, Ritz J, Rivat C, Schambach A, Shaw KL, Sherman EA, Silberstein LE, Six E, Touzot F, Tsytsykova A, Xu-Bayford J, Baum C, Bushman FD, Fischer A, Kohn DB, Filipovich AH, Notarangelo LD, Cavazzana M, Williams DA, Thrasher AJ. A modified gamma-retrovirus vector for X-linked severe combined immunodeficiency. N Engl J Med. 2014 Oct 9;371(15):1407-17. doi: 10.1056/NEJMoa1404588. PMID 25295500